CLINICAL TRIAL: NCT02365675
Title: An Open Randomized Comparative Trial of Four Different Dressings for Cutaneous Coverage in Pemphigus and Pemphigoid
Brief Title: Wound Dressings for Pemphigus and Pemphigoid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Nacional para la Enseñanza y la Investigación de la Dermatología A.C. (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Jose Contreras-Ruiz, Head of the Interdisciplinary Wound and Ostomy Care Center. Division of Dermatology., Hospital General Dr. Manuel Gea González
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-106-2014
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2014-09

CONDITIONS: Pemphigus; Pemphigoid
Keywords: Pemphigus; Pemphigoid; Wound Healing; Itch; Pain; Wound dressing; Topical treatment
MeSH Terms: conditions — Pemphigus; Pemphigoid, Bullous; Pruritus; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cotton gauze with petrolatum (Active Comparator): The dressing to be used is regular cotton gauze impregnated in petrolatum (a mixture of solid hydrocarbons) creating a film that reduces the adherence of the gauze to the wound.
  Interventions: Device: Cotton gauze with petrolatum
- Cellulose acetate with petrolatum (Active Comparator): The dressing to be used is a mesh or tulle base of cellulose acetate polymers that do not easily adhere to the wound impregnated in petrolatum (a mixture of solid hydrocarbons).
  Interventions: Device: Cellulose acetate with petrolatum
- Nanocrystalline silver (Active Comparator): The dressing to be used consists of two layers of a silver-coated, high-density polyethylene mesh, enclosing a single layer of an apertured non-woven fabric of rayon and polyester. The three components are ultrasonically welded together to maintain the integrity of the dressing in use. Silver is applied to the polyethylene mesh by a vapour deposition process, which results in the formation of microscopic 'nanocrystals' of metallic silver.
  Interventions: Device: Nanocrystalline silver (Acticoat)
- Carboxymethylcellulose with ionic silver (Active Comparator): The dressing to be used is a soft, sterile, non- woven pad dressing made from sodium carboxymethylcellulose containing 1.2% silver in an ionic form.
  Interventions: Device: Carboxymethylcellulose with ionic silver (Aquacel Ag)

INTERVENTIONS:
Device: Cotton gauze with petrolatum
  Arms: Cotton gauze with petrolatum
Device: Cellulose acetate with petrolatum
  Other Names: Curity non-adhering dressing
  Arms: Cellulose acetate with petrolatum
Device: Nanocrystalline silver (Acticoat)
  Other Names: Acticoat
  Arms: Nanocrystalline silver
Device: Carboxymethylcellulose with ionic silver (Aquacel Ag)
  Other Names: Aquacel Ag
  Arms: Carboxymethylcellulose with ionic silver

SUMMARY:
The purpose of this study is to compare the efficacy of four dressings (covers) namely: gauze with petrolatum , cellulose acetate with petrolatum , pure carboxymethylcellulose with silver and nanocrystalline silver to improve the new growth of skin, reduce pain and itch in persons suffering from pemphigus and pemphigoid.

DETAILED DESCRIPTION:
Pemphigus and pemphigoid are the most frequently autoinmune bullous diseases seen in dermatology. Despite all the treatments that have been studied for the management of bullous skin diseases, there is insufficient information about the best skin dressing or cover that can be used in affected or denuded areas in these conditions.

Therefore we will compare the efficacy of four different covers (gauze with petrolatum , cellulose acetate with petrolatum , pure carboxymethylcellulose with silver and nanocrystalline silver) in providing faster healing and decreasing pain and itch.

Each patient with the diagnosis of either pemphigus or pemphigoid will have a full skin examination and 4 of the most affected areas will be randomly assigned to receive each of the 4 treatments previously described.

There is no clinical study focused specifically on the materials that will be used in this study. There are few isolated cases reported that can not be taken as a basis. Considering the above and based on the clinical experience, we consider it appropriate to conduct a pilot study with a total of 10-14 patients, with it we will perform a sample calculation, considering a potential alpha error of 0.05, yielding the beta error by subtracting 1.0 to the power sample calculated .

In all of the patients 4 affected areas of 8 cm x 8 cm ( 64 cm2 ) will be selected and marked with the letters A, B , C and D. The investigator will generate randomization tables where previously established and numbered treatments 1 to 4 will be randomly assigned to each of the four areas. Thus all patients will receive the 4 therapies but randomly in the 4 areas previously selected.

The variables that will be studied are:

* Total area affected : Consists of the sum of the percentages of skin that is not healthy in the 64 cm2
* Intensity of pain: sensory unpleasant emotional experience that occurs from the potential or actual injury tissue . Will be assessed by visual analog scale, validated method.
* Erythema: Inflammation of the skin surface caused by excess blood supply, causing redness.
* Itch: cutaneous unpleasant sensation and of variable intensity that causes an urge to scratch to get relief. Will be assessed by visual analog scale, validated method.
* Healing: Reparing process of an altered tissue, resulting in the formation of a scar tissue. Will be measured based on the reduction of wound area percentage. It shall be measured in cm2 with ImageJ® program ( ImageJ® , US National Institutes of Health , Bethesda , Maryland , USA , ( http : //imagej.nih.gov/ij/ ) ) .
* Ulcer: injury depressed by loss of epidermis, dermis and subcutaneous tissue . They will be measured in total area in cm2 by ImageJ® program.
* Blisters, pustules or vesicles: are elemental skin lesions with a liquid content ranging from light to heavy white. They will be measured in total area in cm2 by ImageJ® program.

Procedure description:

Day 0

* The patient will be evaluated to determine if is eligible according to the selection criteria.
* The protocol will be explained in clear words so that the patient understands it.
* The patient will have to sign the informed consent.
* Total body surface area will be revalutatd to select the 4 most severely affected areas in the trunk or limbs of 8 cm x 8 cm each and that will be assigned with a letter from A to D.
* With an indelible marker the 4 vertices of each of the previously selected areas will be marked.
* A label graduated in millimeters will be placed at the bottom edge of the marked areas.
* A panoramic picture of each of the four areas will be taken to ensure that if the label is lost, we can replicate it in the next visit.
* An aproach picture of each of these four areas will be taken.
* The selected areas will be cleaned with sterile saline.
* Clinical evaluation will be performed and the section of the report format will be filled.
* The envelope containing randomization numbers will be opened to decide which dressing skin cover will be used to each of the selected areas.
* The dressings (covers) will be placed on each of the selected areas. Above it conventional gauze will be placed and this cure will be pinned up with conventional elastic white band.
* The patient will recieve the appointments of the 6 subsequent valorations.
* The patient will recive the prescription for the systemic management of the bullous skin disease.
* The patient will receive a second prescription explaining how he should be healing between each visit. If it is an inpatient, the healing and measurement will be performed by the medical personnel assigned. The family will be explained how to perform the healing and at the end of his hospital stay a prescription will be given with the instructions. Also the next control appointment will be given.
* Pictures will be downloaded and the presence of abnormal skin will be measured using a standardized measurement program ( ImageJ® , US NationalInstitutes of Health , Bethesda , Maryland , USA , ( http://imagej.nih.gov/ij/ ) ). All data obtained will be registered in the report format made specifically for this trial.

Subsequent visits ( 7, 14, 21 , 28, 35 )

* The presence of systemic or local adverse effects at any of the 4 areas of study will be asked.
* The 4 areas will be discovered using saline and gently drying. The healling and the further steps are the same as the ones explained above.
* All the data obtained will be recorded on the report format.

Final visit (day 42)

* The patient will be told he or she is no more in the protocol and which of the dressings worked the best.
* The patient will receive his or her next appoinment.
* A prescription with the systemic treatment will be given.
* A second prescription will be given, explaining how to perform the healings.
* All data obtained will be recorded to the further results analysis.

Results will be presented as percentages or proportions for categorical variables and by mean ± standard deviation for continuous variables. The percentage of epithelialization between the four groups will be compared with Chi Square RxC. Continuous numerical variables will be compared with one way ANOVA in the case of homoscedastic variances or by Kruskall Wallis variance in the case of heteroskedastic variances. The results will be adjusted in relation to the received systemic treatment (duration, intensity), the location of the lesions and its chronicity with multivariate lienal regression analysis . For bivariate anaysis a significant value of p < 0.05 will be used. For multivariate analysis a p < 0.10 value will be used. STATA version 13.0 for Mac wiil be used.

Tables and grapfhs will be used to present the results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pemphigus vulgaris, pemphigus foliaceus , pemphigus vegetans, paraneoplastic pemphigus or bullous pemphigoid
* At least four areas of active disease in the trunk or limbs of 8 x 8 cm characterized by denudation, ulceration, scabs or blisters.
* Capable of being evaluated weekly either as outpatient or hospitalized
* Actively treated with immunosuppressive or immunomodulatory drugs for pemphigus or pemphigoid control
* Willing to sign an informed consent

Exclusion Criteria:

* Patients with hypersensitivity to any of the components of the skin dressings that will be used.
* Patients who have participated in any clinical trial in the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Wound Healing Percentage of a 64 cm2 area of epithelialized skin | 42 days
  Percentage of a 64 cm2 area of epithelialized skin

SECONDARY OUTCOMES:
Pain Using the visual analog scale a decrease in pain score | 42 days
  Using the visual analog scale a decrease in pain score
Itch Using the visual analog scale a decrease in itch score | 42 days
  Using the visual analog scale a decrease in itch score

CONTACTS AND LOCATIONS:
Overall Officials: Jose Contreras-Ruiz, MD, Principal Investigator — Hospital General Dr Manuel Gea Gonzalez
Locations (2):
- Mexico (2):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Hospital General Dr Manuel Gea González, Mexico City, Mexico City

REFERENCES:
- [Background] Amagai M. Preface to Journal of Dermatology special issue: pemphigus updates from around the world. J Dermatol. 2015 Jan;42(1):2. doi: 10.1111/1346-8138.12774. No abstract available. PMID 25558945
- [Background] Mimouni D, Anhalt GJ, Lazarova Z, Aho S, Kazerounian S, Kouba DJ, Mascaro JM Jr, Nousari HC. Paraneoplastic pemphigus in children and adolescents. Br J Dermatol. 2002 Oct;147(4):725-32. doi: 10.1046/j.1365-2133.2002.04992.x. PMID 12366419
- [Background] Mutasim DF. Autoimmune bullous dermatoses in the elderly: an update on pathophysiology, diagnosis and management. Drugs Aging. 2010 Jan 1;27(1):1-19. doi: 10.2165/11318600-000000000-00000. PMID 20030429
- [Background] Kirtschig G, Khumalo NP. Management of bullous pemphigoid: recommendations for immunomodulatory treatments. Am J Clin Dermatol. 2004;5(5):319-26. doi: 10.2165/00128071-200405050-00005. PMID 15554733
- [Background] Martin LK, Werth V, Villanueva E, Segall J, Murrell DF. Interventions for pemphigus vulgaris and pemphigus foliaceus. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD006263. doi: 10.1002/14651858.CD006263.pub2. PMID 19160272
- [Background] Joly P, Roujeau JC, Benichou J, Delaporte E, D'Incan M, Dreno B, Bedane C, Sparsa A, Gorin I, Picard C, Tancrede-Bohin E, Sassolas B, Lok C, Guillaume JC, Doutre MS, Richard MA, Caux F, Prost C, Plantin P, Chosidow O, Pauwels C, Maillard H, Saiag P, Descamps V, Chevrant-Breton J, Dereure O, Hellot MF, Esteve E, Bernard P. A comparison of two regimens of topical corticosteroids in the treatment of patients with bullous pemphigoid: a multicenter randomized study. J Invest Dermatol. 2009 Jul;129(7):1681-7. doi: 10.1038/jid.2008.412. Epub 2009 Jan 29. PMID 19177141
- [Background] Wojnarowska F, Kirtschig G, Highet AS, Venning VA, Khumalo NP; British Association of Dermatologists. Guidelines for the management of bullous pemphigoid. Br J Dermatol. 2002 Aug;147(2):214-21. doi: 10.1046/j.1365-2133.2002.04835.x. PMID 12174090
- [Background] Khumalo NP, Murrell DF, Wojnarowska F, Kirtschig G. A systematic review of treatments for bullous pemphigoid. Arch Dermatol. 2002 Mar;138(3):385-9. doi: 10.1001/archderm.138.3.385. PMID 11902990
- [Background] Kirtschig G, Middleton P, Bennett C, Murrell DF, Wojnarowska F, Khumalo NP. Interventions for bullous pemphigoid. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD002292. doi: 10.1002/14651858.CD002292.pub3. PMID 20927731
- [Background] Dressler DP, Skornik WA. Burn wound dressings. II. Effect on wound sepsis. J Trauma. 1971 Apr;11(4):325-30. No abstract available. PMID 5551730
- [Background] Sibbald RG, Contreras-Ruiz J, Coutts P, Fierheller M, Rothman A, Woo K. Bacteriology, inflammation, and healing: a study of nanocrystalline silver dressings in chronic venous leg ulcers. Adv Skin Wound Care. 2007 Oct;20(10):549-58. doi: 10.1097/01.ASW.0000294757.05049.85. PMID 17906429
- [Background] Gravante G, Caruso R, Sorge R, Nicoli F, Gentile P, Cervelli V. Nanocrystalline silver: a systematic review of randomized trials conducted on burned patients and an evidence-based assessment of potential advantages over older silver formulations. Ann Plast Surg. 2009 Aug;63(2):201-5. doi: 10.1097/SAP.0b013e3181893825. PMID 19571738
- [Background] Asz J, Asz D, Moushey R, Seigel J, Mallory SB, Foglia RP. Treatment of toxic epidermal necrolysis in a pediatric patient with a nanocrystalline silver dressing. J Pediatr Surg. 2006 Dec;41(12):e9-12. doi: 10.1016/j.jpedsurg.2006.08.043. PMID 17161178
- [Background] Chen J, Han CM, Lin XW, Tang ZJ, Su SJ. [Effect of silver nanoparticle dressing on second degree burn wound]. Zhonghua Wai Ke Za Zhi. 2006 Jan 1;44(1):50-2. Chinese. PMID 16620649
- [Background] Murrell DF, Daniel BS, Joly P, Borradori L, Amagai M, Hashimoto T, Caux F, Marinovic B, Sinha AA, Hertl M, Bernard P, Sirois D, Cianchini G, Fairley JA, Jonkman MF, Pandya AG, Rubenstein D, Zillikens D, Payne AS, Woodley D, Zambruno G, Aoki V, Pincelli C, Diaz L, Hall RP, Meurer M, Mascaro JM Jr, Schmidt E, Shimizu H, Zone J, Swerlick R, Mimouni D, Culton D, Lipozencic J, Bince B, Grando SA, Bystryn JC, Werth VP. Definitions and outcome measures for bullous pemphigoid: recommendations by an international panel of experts. J Am Acad Dermatol. 2012 Mar;66(3):479-85. doi: 10.1016/j.jaad.2011.06.032. Epub 2011 Nov 5. PMID 22056920
- [Background] Daroczy J, Szalai I. [Use of polyurethane foil for wound covering]. Orv Hetil. 1991 Jun 2;132(22):1203-4. Hungarian. PMID 2067830
- [Background] Patange VS, Fernandez RJ, Motla MU, Mahajan SA. Dressing wounds with potato peel. Indian J Dermatol Venereol Leprol. 1996 Sep-Oct;62(5):286-8. PMID 20948091
- [Background] Dumas V, Roujeau JC, Wolkenstein P, Revuz J, Cosnes A. The treatment of mild pemphigus vulgaris and pemphigus foliaceus with a topical corticosteroid. Br J Dermatol. 1999 Jun;140(6):1127-9. doi: 10.1046/j.1365-2133.1999.02895.x. PMID 10354082
- [Background] Grando SA. New approaches to the treatment of pemphigus. J Investig Dermatol Symp Proc. 2004 Jan;9(1):84-91. doi: 10.1111/j.1087-0024.2004.00826.x. PMID 14870992
- [Background] Vun YY, Lun K, Strutton G. Use of biosynthetic dressings in paraneoplastic pemphigus. Australas J Dermatol. 2004 May;45(2):133-5. doi: 10.1111/j.1440-0960.2004.00067.x. PMID 15068464